CLINICAL TRIAL: NCT00692731
Title: A Randomized, Double-Blind, Controlled Study to Assess the Efficacy of a Tea Catechin Sports Drink for Enhancing Exercise-Induced Fat Loss
Brief Title: Efficacy of a Tea Catechin Sports Drink for Enhancing Exercise-Induced Fat Loss
Status: Completed | Type: Observational
Sponsor: Provident Clinical Research (Other)
Collaborators: Kao (Taiwan) Corporation (Industry)
Responsible Party: Kevin C. Maki, PhD, Provident Clinical Research
Other Study IDs: PRV-06001
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Overweight; Obesity
Keywords: green tea,; polyphenols,; weight loss,; body fat
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Catechin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active: Tea catechin sport beverage
  Interventions: Dietary Supplement: 500 mL/day of a beverage providing approximately 625 mg catechins
- Control: Control beverage
  Interventions: Other: Control beverage matched for energy and caffeine content

INTERVENTIONS:
Dietary Supplement: 500 mL/day of a beverage providing approximately 625 mg catechins — Subjects were asked to consume 500 mL/day of a beverage providing approximately 625 mg catechins
  Groups: Active
Other: Control beverage matched for energy and caffeine content — 500 mL/day of a control beverage
  Groups: Control

SUMMARY:
The primary objective of this trial is to evaluate the influence of consuming a tea catechin containing sports beverage on body fat mass during exercise-induced weight loss among overweight and obese men and women.

DETAILED DESCRIPTION:
The study will include two screening/baseline visits and six treatment visits over 12 weeks. During the treatment phase of the study, subjects will be instructed to consume one bottle of sports drink (500 ml) daily (total consumption of tea catechins in the active group = 540 mg/d). Subjects will be asked to maintain a constant energy intake throughout the study period. Three-day diet records will be collected and analyzed at weeks 0, 6, and 12 to evaluate consistency of energy intake.

All subjects will engage in an exercise program with a goal of maintaining 180 min/week of low- to moderate-intensity exercise (e.g., walking and other aerobic activities, 4-6 days per week). Three of the weekly exercise sessions will be supervised and 1-3 will be unsupervised. Subjects will be asked to wear a pedometer and record their daily physical activity (steps) each night in a physical activity diary. Diaries will be collected at each visit and used to evaluate exercise compliance. Dual energy X-ray absorptiometry (DEXA) and computed tomography (CT) scans will be performed at baseline (week 0) and at the end of the treatment (week 12). Additionally, body weight and abdominal circumference will be assessed at every clinic visit during the study. It is anticipated that subjects will expend 1000-1800 kcal per week above their baseline level in deliberate physical activity. Accordingly, the control group is expected to lose 1.5 to 2.8 kg of body fat during the 12-week treatment period

ELIGIBILITY:
Inclusion Criteria:

* Men and women 21 to 65 years of age, inclusive
* Waist circumference ≥ 87 cm for women and ≥ 90 cm for men at screening
* Total cholesterol ≥ 200 mg/dL
* Provide written informed consent and authorization for protected health information

Exclusion Criteria:

* Volunteers with Body mass index ≥ 40.0 kg/m2 or < 25.0 kg/m2;
* Recent weight loss of more than 4.5 kg;
* Recent use of any weight loss medications, supplements, or programs;
* History of weight-reducing surgery or an eating disorder
* Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects included generally healthy, normally sedentary men and women. Eligible participants were required to be 21 to 65 years of age, have a waist circumference ≥ 87 cm (women) or ≥ 90 cm (men), and total cholesterol ≥ 200 mg/dL at screening.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Changes in body fat mass. | Baseline to end-of-treatment

SECONDARY OUTCOMES:
Changes in body weight | Baseline to end-of-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — Provident Clinical Research
Locations (2):
- United States (2):
  - Meridien Research, St. Petersburg, Florida
  - Provident Clinical Research, Bloomington, Indiana

REFERENCES:
- [Background] Murase T, Nagasawa A, Suzuki J, Hase T, Tokimitsu I. Beneficial effects of tea catechins on diet-induced obesity: stimulation of lipid catabolism in the liver. Int J Obes Relat Metab Disord. 2002 Nov;26(11):1459-64. doi: 10.1038/sj.ijo.0802141. PMID 12439647
- [Background] Dulloo AG, Duret C, Rohrer D, Girardier L, Mensi N, Fathi M, Chantre P, Vandermander J. Efficacy of a green tea extract rich in catechin polyphenols and caffeine in increasing 24-h energy expenditure and fat oxidation in humans. Am J Clin Nutr. 1999 Dec;70(6):1040-5. doi: 10.1093/ajcn/70.6.1040. PMID 10584049
- [Background] Nagao T, Komine Y, Soga S, Meguro S, Hase T, Tanaka Y, Tokimitsu I. Ingestion of a tea rich in catechins leads to a reduction in body fat and malondialdehyde-modified LDL in men. Am J Clin Nutr. 2005 Jan;81(1):122-9. doi: 10.1093/ajcn/81.1.122. PMID 15640470
- [Background] Nagao T, Hase T, Tokimitsu I. A green tea extract high in catechins reduces body fat and cardiovascular risks in humans. Obesity (Silver Spring). 2007 Jun;15(6):1473-83. doi: 10.1038/oby.2007.176. PMID 17557985